CLINICAL TRIAL: NCT04943757
Title: Graft-versus-host Disease Prophylaxis With Combination of Post-transplantation Benadamustine and Cyclophosphamide in Patients With Refractory Myeloid Malignancies (PTBCy)
Brief Title: Post-transplantation Benadamustine and Cyclophosphamide in Patients With Refractory Myeloid Malignancies
Acronym: PTBCy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Principal Investigator, Ivan S Moiseev, Vice-director for science RM Gorbacheva Institute, St. Petersburg State Pavlov Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05/21-n
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Myeloid Leukemia, Acute; Chronic Myeloid Leukemia; Myelodysplastic Syndromes; Myeloproliferative Neoplasm
Keywords: Bendamustine; Cyclophosphamide; Graft-versus-host disease; Graft-versus-leukemia effect; Refractory; Acute Myeloid leukemia; Hematopoietic Stem Cell Transplantation; Allogeneic
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Myeloproliferative Disorders; Graft vs Host Disease | interventions — Bendamustine Hydrochloride; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PTBCy graft-versus-host disease prophylaxis (Experimental): Days +3 through +4: Bendamustine 50 mg/m2 iv x 2 days; Days +3 through +4: Cyclophosphamide 25 mg/kg iv x 2 days; Days +5 through +35: Mycophenolate mofetil 30 mg/kg/day, maximum 3 g/day, iv or po x 30 days; Days +5 through +100: Tacrolimus 0.03 mg/kg/day with further correction by concentration
  Interventions: Drug: Bendamustine Hydrochloride; Drug: Cyclophosphamid

INTERVENTIONS:
Drug: Bendamustine Hydrochloride — 50 mg/m2 iv Days +3 through +4 after allogeneic hematopoietic stem cell transplantation
Drug: Cyclophosphamid — 25 mg/kg iv Days +3 through +4 after allogeneic hematopoietic stem cell transplantation

SUMMARY:
Prognosis of patients undergoing salvage allogeneic stem cell transplantation for refractory leukemia or other refractory myeloid malignanies is poor. One of the approaches to augment graft-versus-leukemia effect the use of post-transplantation bendamustine in graft-versus-host disease prophylaxis. Despite high frequency of responses and durable remissions after this approach majority of patients develop a serious complication - cytokine release syndrome, which can be life-threatening in some patients. On the other hand post-transplantation cyclophocphamide was reported to abort cytokine release syndrome that sometimes occurs after graft transfusion in patients after haploidentical graft transfusion. The aim of this study is to evaluate if the combination of post-transplantation bendamustine (PTB) and post-transplantation cyclophosphamide (PTCY) facilitates comparable graft-versus leukemia effect to PTB, but with better safety profile and reduced incidence of severe cytokine release syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with indication for allogeneic hematopoietic stem cell transplantation
* Patients with 5-10/10 HLA-matched related or unrelated donor available. The donor and recipient must be identical by the following genetic loci: HLA-A, HLA-B, HLA-Cw, HLA-DRB1, and HLA-DQB1.
* Peripheral blood stem cells or bone marrow as a graft source
* Diagnosis:

Acute myeloid leukemia Chronic myeloid leukemia, Ph+ Myelodysplastic Syndromes Myeloprolipherative neoplasms

* Salvage hematopoietic stem cell transplantation defined as:
* Acute myeloid leukemia: >5% of clonal blasts despite adequate previous induction therapy or allogeneic stem cell transplantation Myelodysplastic Syndrome: >10% of blasts despite previous therapy with -7 or complex karyotype, or p53 mutation Chronic myeloid leukemia: blast crisis or acceleration phase despite at least 3 previous lines of TKIs Myeloprolipherative neoplasms : high tumor burden despite previous therapy, including >20 000 WBC/ ul or splenomegaly >15 cm
* No severe concurrent illness

Exclusion Criteria:

* Moderate or severe cardiac dysfunction, left ventricular ejection fraction <50%
* Moderate or severe decrease in pulmonary function, FEV1 <70% or DLCO<70% of predicted
* Respiratory distress >grade I
* Severe organ dysfunction: AST or ALT >5 upper normal limits, bilirubin >1.5 upper normal limits, creatinine >2 upper normal limits
* Creatinine clearance < 60 mL/min
* Uncontrolled bacterial or fungal infection at the time of enrollment
* Requirement for vasopressor support at the time of enrollment
* Karnofsky index <30%
* Pregnancy
* Somatic or psychiatric disorder making the patient unable to sign informed consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-05-30 (Actual)

PRIMARY OUTCOMES:
Event-free survival analysis [ Time Frame: 1 year ] | 1 year
  Measure: Kaplan-Meier estimate of death or relapse, or graft failure

SECONDARY OUTCOMES:
- Incidence of Cytokine release syndrome | 100 days
  Proportion of patients with cytokine release syndrome according to ASBMT Consensus Grading for Cytokine Release Syndrome, 2018
Incidence of HSCT-associated adverse events (safety and toxicity) | 100 days
  Toxicity assessment is based on NCI CTC AE 5.0 grades. Veno-occlusive disease incidence and severity assessment is based on EBMT criteria 2016. Transplant-associated microangiopathy incidence assessment is based on Cho et al.
Incidence of acute GVHD grade II-IV | 125 days
  Cumulative incidence of patients with acute GVHD II-IV grade
Incidence of moderate and severe chronic GVHD | 1 year
  Cumulative incidence of patients with moderate and severe chronic GVHD according to NIH 2015 criteria
Relapse rate analysis | 1 year
  Cumulative incidence of patients with relapse
Non-relapse mortality analysis | 1 year
  Cumulative incidence of patients with mortality without hematological relapse of malignancy
Overall survival analysis | 1 year
  Kaplan-Meier estimate of death from all causes

CONTACTS AND LOCATIONS:
Locations (1):
- RM Gorbacheva Research Institute, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Yes
Request for sharing data with the study plan for the data will be evaluated under common conditions by Pavlov University Ethical Committee.

REFERENCES:
- [Background] Moiseev I, Bondarenko S, Morozova E, Vlasova Y, Dotsenko A, Epifanovskaya O, Babenko E, Botina A, Baykov V, Surkova E, Lapin S, Beynarovich A, Borzenkova E, Golosgchapov O, Kanunnikov M, Kudyasheva O, Ovechkina V, Pirogova O, Porunova V, Rudakova T, Smikova O, Smirnova A, Afansyev B. Graft-versus-Host Disease Prophylaxis with Post-Transplantation Bendamustine in Patients with Refractory Acute Leukemia: A Dose-Ranging Study. Transplant Cell Ther. 2021 Jul;27(7):601.e1-601.e7. doi: 10.1016/j.jtct.2021.03.032. Epub 2021 May 7. PMID 33845259